CLINICAL TRIAL: NCT05052567
Title: Phase 1b/2 Clinical Study on Safety, Pharmacokinetics, and Preliminary Efficacy of CEND-1 for Injection in Patients With Advanced Metastatic Pancreatic Ductal Adenocarcinoma
Brief Title: CEND-1 Injection (QLC12102) in Patients With Advanced Metastatic Pancreatic Ductal Adenocarcinoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Collaborators: Cend Therapeutics Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CEND1-201
Record Dates: First submitted 2021-08-29; First posted 2021-09-22 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2022-01

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CEND-1 (Experimental): CEND-1+paclitaxel (albumin-bound type)+gemcitabine
  Interventions: Drug: CEND-1

INTERVENTIONS:
Drug: CEND-1 — The dose is specified according to the protocol. CEND-1+paclitaxel (albumin-bound type)+gemcitabine
  Other Names: iRGD; LSTA1; certepetide

SUMMARY:
The purpose of this study was to evaluate the preliminary safety, efficacy and PK characteristics of cend-1 in patients with advanced metastatic pancreatic ductal adenocarcinoma (Chinese population).

DETAILED DESCRIPTION:
This study is a multi-center, non-randomized, open-label phase Ib/II clinical study carried out in Chinese patients with advanced metastatic pancreatic ductal adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 to 80 years old, male or female.
* Patients with histologically confirmed metastatic pancreatic ductal adenocarcinoma;
* The Eastern Cooperative Oncology Group (ECOG) score is 0 to 1.
* The life expectancy is no less than 12 weeks.
* According to the RECIST v1.1 evaluation criteria, the patient has at least one measurable lesion (exclude if there is only a target lesion located at a site previously treated with radiation);
* The patient who is suitable for first-line treatment with a combined regimen of paclitaxel (albumin-bound type) and gemcitabine;

Exclusion Criteria:

* The patients who have been previously treated with chemotherapy or other drugs for pancreatic carcinoma, or who have been treated with other anti-cancer drugs, including chemotherapy, targeted therapy, immunotherapy, or biologics.
* The patients who are known to be allergic to the investigatinal drug (CEND-1 analogue) or its any excipient;
* The patients with the following conditions: myocardial infarction, severe/unstable angina, NYHA grade 2 or above cardiac dysfunction, and clinically significant supraventricular or ventricular arrhythmia requiring clinical intervention within 6 months before signing the ICF;
* The patients with symptomatic CNS metastasis, leptomeningeal metastases, or spinal cord compression due to metastasis. However, the patients with symptomatic CNS metastasis before first administration of the investigational drug, who is treated and stable for no less than 4 weeks, and the systematic hormone (any dose) treatment has been stopped for over 2 weeks, can be enrolled;
* The patients with other active malignant tumors within 3 years before signing the ICF. The cured skin basal cell carcinoma or squamous cell carcinoma, superficial bladder cancer, carcinoma in situ of the cervix, carcinoma in situ of the breast ductal, and papillary thyroid cancer are excluded.
* The patients with human immunodeficiency virus (HIV) infection or known acquired immunodeficiency syndrome (AIDS), active hepatitis or co-infection with hepatitis B and C.
* The patients who participated in any other drug clinical trial and administrated the investigational drug within 4 weeks before first dose;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-10-21 (Actual); Primary Completion 2024-06-29 (Actual); Study Completion 2024-06-29 (Actual)

PRIMARY OUTCOMES:
Safety of CEND-1 mesured by AEs, SAEs and treatment related adverse events. | 12 month
  Adverse events (AEs), serious adverse events (SAEs), treatment related adverse events are included. The investigator should carry out judgment for investigational drug correlation.
Preliminary efficacy of CEND-1 mesured by ORR, DOR, DCR, OS, PFS ect. | 12 month
  Objective response rate (ORR), duration of response (DOR), disease control rate (DCR), overall survival (OS), progress-free survival (PFS), PFS rate, OS rate etc. are included.

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China